CLINICAL TRIAL: NCT06851975
Title: Research Into Biomarkers Predictive of Survival and Response to Cancer Treatment
Acronym: BEST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018-61
Record Dates: First submitted 2025-02-14; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- principal (Other): blood sampling
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — 36ml of blood will be taken during a blood sampling performed in standard practice

SUMMARY:
Research into biomarkers predictive of survival and response to cancer treatment

ELIGIBILITY:
Inclusion Criteria:

* Patient having a blood test, venous line insertion or injection on an implantable venous device scheduled as part of their standard care,
* Patient who has read the information note and stated that he/she has no objections
* Patient who has not objected to the use of this data for medical research purposes
* Patient with social security cover.

Exclusion Criteria:

* Patient already included in the study
* Patient considered to be a vulnerable person; vulnerable persons are defined in article L1121-5 to -8

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40000 (Estimated)
Dates: Start 2020-01-07 (Actual); Primary Completion 2099-12-31 (Estimated); Study Completion 2099-12-31 (Estimated)

PRIMARY OUTCOMES:
Prediction | day 1
  The aim of this project is to make a biobank in prevision of MR004 sub-projects which define specific biomarkers studied to identify biomarkers predictive of response.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Antoine Lacassagne, Nice, France

IPD SHARING:
Plan to Share IPD: Yes
pseudonymised data will only be collected
Supporting Information: Study Protocol, CSR
Time Frame: at the end of study